CLINICAL TRIAL: NCT06194786
Title: Diet and Physical Activity Program in Colorectal Cancer Survivor: a Randomized Controlled Trial
Acronym: DPAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Habib Bourguiba University Hospital (Other)
Collaborators: National cancer institute -Misurata (Unknown)
Responsible Party: Principal Investigator, Wala Ben Kridis, Principal Investigator, Habib Bourguiba University Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 04/2023
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Colorectal Cancer
Keywords: Diet; Physical activity
MeSH Terms: conditions — Colorectal Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Dietary and physical activity
  Interventions: Behavioral: Group D
- Group B (Experimental): Dietary only
  Interventions: Behavioral: Group D
- Group C (Experimental): Physical activity only
  Interventions: Behavioral: Group D

INTERVENTIONS:
Behavioral: Group D — Usual care

SUMMARY:
Colorectal cancers (CRC) represent the 1st digestive cancer and the 3rd cancer in the world. The World Cancer Research Fund summarized evidence from observational studies and concluded that low dietary fiber, and high red and processed meat (RPM) intakes were associated with higher risk of (CRC), whilst physical activity (PA) protected against developing colon cancer.

Post-treatment management is essential for improving the health and quality of life of colorectal cancer (CRC) survivors. The number of cancer survivors is continually increasing, which is causing a corresponding growth in the need for effective post- treatment management programs. To date, there is insufficient information available from the published literature as to the most effective way in promoting lifestyle changes in CRC survivors. Moreover, none of these interventions have been conducted in an African population. We aim to assess whether the proposed program may effectively modify the targeted behaviors, to evaluate whether the dietary and PA interventions of the "Moving Bright, Eating Smart" program are effective in reducing the consumption of red and processed meat (RPM) and refined grain (RG), increasing the physical activity (PA) levels in north African (Libyan and Tunisian) adult colorectal cancer (CRC) survivors and to assess the efficacy of behavioral interventions on cancer outcomes (overall survival, disease free survival).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven colorectal adenocarcinoma patients above the age of 18 years within one year of completion of main cancer treatment who are able to provide informed consent.

Exclusion Criteria:

* Colorectal cancer patients who have persistent or recurrent disease at the time of the recruitment, are receiving cancer treatment, have known contraindication to physical activity, have psychiatric disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
physical activity target-cancer outcome | 0-6-12-18-24 months
  accelerometer or stopwatch or phone timer
Dietary target-red meat | 0-6-12-18-24 months
  food frequency questionnaire

SECONDARY OUTCOMES:
overall survival | 12-2 months
  time between randomization and date of last news
Disease free survival | 12-24 months
  time between randomization and progression

CONTACTS AND LOCATIONS:
Locations (1):
- Wala Ben Kridis, Sfax, Tunisia

REFERENCES:
- [Derived] Aboturkia AM, Ben Kridis W, Aqoup MO, Abdoalmola MO, Ben Ali S, Khanfir A. Diet and physical activity in colorectal cancer patients: A research protocol of a randomized controlled study. World J Gastrointest Oncol. 2025 Aug 15;17(8):109579. doi: 10.4251/wjgo.v17.i8.109579. PMID 40837756